CLINICAL TRIAL: NCT03129139
Title: A Phase 1, Multi-Center, Open-Label, Dose-Escalation, Safety, Pharmacokinetic, and Pharmacodynamic Study of Minnelide™ Capsules Given Alone or in Combination With Protein-Bound Paclitaxel in Patients With Advanced Solid Tumors
Acronym: Minnelide 101
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Minneamrita Therapeutics LLC (Industry)
Collaborators: Translational Drug Development (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Minnelide 101
Record Dates: First submitted 2017-04-18; First posted 2017-04-26 (Actual); Last update posted 2023-10-18 (Actual); Status verified 2023-10

CONDITIONS: Advanced Cancer; Gastric Cancer; Breast Cancer; Pancreatic Cancer; Prostate Cancer Metastatic; Colo-rectal Cancer; Solid Tumor; Solid Carcinoma; Solid Carcinoma of Stomach; Cancer of Stomach
Keywords: Metastatic
MeSH Terms: conditions — Stomach Neoplasms; Breast Neoplasms; Pancreatic Neoplasms; Colonic Neoplasms; Neoplasm Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Regimen A (monotherapy) (Experimental): Minnelide™ Capsules will be given as a single agent orally once daily x 21 days followed by a 7-day off schedule. One cycle will equal 28 days. MinnelideTM Capsules should be given with the patient in a fasting state.
  Interventions: Drug: Minnelide™Capsules
- Regimen B (combination) (Experimental): MinnelideTM Capsules will be given orally once daily x 21 days in combination with protein-bound paclitaxel given intravenously on days 1, 8 and 15 in patients with pancreas and breast cancer. One cycle will equal 28 days. MinnelideTM Capsules should be given with the patient in a fasting state.
  Interventions: Drug: Minnelide™Capsules
- Regimen C (monotherapy in Gastric Cancer) (Experimental): Minnelide™ Capsules will be given as a single agent orally once daily x 21 days followed by a 7-day rest period. One cycle will equal 28 days. Minnelide™ Capsules should be given with the patient in a fasting state.
  Interventions: Drug: Minnelide™Capsules

INTERVENTIONS:
Drug: Minnelide™Capsules — Minnelide™ is a water soluble disodium salt variant of triptolide an heat shock protein (HSP) inhibitor.

SUMMARY:
A Phase I, Multicenter, Open-label, Dose-Escalation, Safety, Pharmacokinetic and Pharmacodynamic Study of Minnelide™Capsules given daily for 21 days followed by 7 days off schedule in patients with Advanced Solid Tumors

ELIGIBILITY:
Inclusion:

* Patients with histologically confirmed advanced solid tumors (regimen A), breast or pancreas (regimen B), or gastric cancer (regimen C)
* Tumor progression after receiving standard/approved chemotherapy or where there is no approved therapy
* Prior treatment with protein-bound paclitaxel allowed if it has been six months since received or progressed on protein-bound paclitaxel and plan to continue to receive protein-bound paclitaxel with MinnelideTM Capsules
* One or more metastatic tumors measurable per RECIST v1.1 Criteria
* Karnofsky performance ≥ 70%
* Life expectancy of at least 3 months
* Age ≥ 18 years
* Signed, written IRB-approved informed consent
* A negative pregnancy test (if female)
* Acceptable liver function:

  * Bilirubin ≤ 1.5 times upper limit of normal
  * AST (SGOT), ALT (SGPT) and Alkaline phosphatase ≤ 2.5 times upper limit of normal (if liver metastases are present, then ≤ 5 x ULN is allowed)
  * Albumin ≥ 3.0 g/dL
* Acceptable renal function:

  o Serum creatinine within normal limits, OR calculated creatinine clearance ≥ 60 mL/min/1.73 m2 for patients with creatinine levels above institutional normal.
* Acceptable hematologic status:

  * Granulocyte ≥ 1500 cells/mm3
  * Platelet count ≥ 100,000 (plt/mm3)
  * Hemoglobin ≥ 9 g/dL
* Urinalysis:

  o No clinically significant abnormalities
* Acceptable coagulation status:

  * PT ≤ 1.5 times institutional ULN
  * PTT ≤ 1.5 times institutional ULN
* For men and women of child-producing potential, the use of effective contraceptive methods during the study

Exclusion Criteria:

* New York Heart Association Class III or IV, cardiac disease, myocardial infarction within the past 6 months, unstable arrhythmia, or evidence of ischemia on ECG
* Baseline QTc exceeding 470 msec (using the Bazett's formula) and/or patients receiving class 1A or class III antiarrhythmic agents.
* Active, uncontrolled bacterial, viral, or fungal infections, requiring systemic therapy
* Pregnant or nursing women. NOTE: Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; or abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.
* Treatment with radiation therapy, surgery, chemotherapy, or investigational therapy within one month prior to study entry (6 weeks for nitrosoureas or Mitomycin C).
* Unwillingness or inability to comply with procedures required in this protocol
* Known infection with HIV, hepatitis B, or hepatitis C
* Serious nonmalignant disease (e.g., hydronephrosis, liver failure, or other conditions) that could compromise protocol objectives in the opinion of the investigator and/or the sponsor
* Patients who are currently receiving any other investigational agent
* Patients who are on a prohibited medication (section 4.4.2).
* Patients with biliary obstruction and/or biliary stent (Regimen B only)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2017-10-10 (Actual); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Number of Participants With Treatment-Related Adverse Events | 24 months
  as assessed by CTCAE V4 .03
Anti-tumor activity | 24 months
  RECIST 1.1

CONTACTS AND LOCATIONS:
Overall Officials: Jordan Jacobs, MBA, Study Director — Translational Drug Development
Locations (7):
- United States (7):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Mayo Clinic Arizona, Phoenix, Arizona
  - HonorHealth Research Institute, Scottsdale, Arizona
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Mayo Clinic, Jacksonville, Florida
  - Mayo Clinic, Rochester, Minnesota
  - Wake Forest Baptist Health, Winston-Salem, North Carolina

IPD SHARING:
Plan to Share IPD: No